CLINICAL TRIAL: NCT05997498
Title: The Effect of Mechanical Dilatation of the Cervix at Elective Caesarean Section on Post-operative Morbidity
Brief Title: Mechanical Dilatation of the Cervix at Elective Caesarean Section on Post-operative Morbidity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Mechanical Dilatation CS
Record Dates: First submitted 2023-07-26; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Cesarean Section Complications
Keywords: Cesarean Section; Mechanical Dilatation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: A statistician prepared a computer-generated random tableand placed the group allocation in serially numbered closed opaque envelopes in a 1:1 ratio. Packing, sealing and numbering will be performed by two independent doctors other than the investigator.
  Patients are allocated to either study group (cervical dilatation) or control group (no cervical dilatation). Allocation will be never changed after opening the envelopes. All patients are blinded to the allocation to avoid bias.
  Neither the investigator nor the outcome assessor following up the patient postoperatively are aware whether the patient had undergone cervical dilation during the cesarean section or not (double-blinding). Randomization coding tables will be hidden from the investigator till the end of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dilation group (Experimental): mechanical cervical dilatation will be done.
  Interventions: Procedure: mechanical cervical dilatation
- control (No Intervention): in which no mechanical cervical dilatation will be done.

INTERVENTIONS:
Procedure: mechanical cervical dilatation — mechanical cervical dilatation during elective cesarean section
  Arms: dilation group

SUMMARY:
The study aims to evaluate the effects of cervical dilatation during cesarean section on postoperative maternal morbidity through different clinical parameters.

DETAILED DESCRIPTION:
A randomized double-blind clinical trial comparing cervical dilatation during caesarean section to no intervention.

* Study participants and sample size This study will include pregnant women with a singleton fetus at term ≥37 weeks of gestation and will be scheduled for elective caesarean section. Eligible participants will be allocated either to the study group (women with intraoperative cervical dilatation) or the control group (women with no intraoperative cervical dilatation).
* Types of interventions Mechanical dilatation of the cervix using a finger, sponge forceps during non-labour caesarean section ***Randomization and Allocation A statistician prepared a computer-generated random tableand placed the group allocation in serially numbered closed opaque envelopes in a 1:1 ratio. Packing, sealing and numbering will be performed by two independent doctors other than the investigator.

Patients are allocated to either study group (cervical dilatation) or control group (no cervical dilatation). Allocation will be never changed after opening the envelopes. All patients are blinded to the allocation to avoid bias.

**Neither the investigator nor the outcome assessor following up the patient postoperatively are aware whether the patient had undergone cervical dilation during the cesarean section or not (double-blinding). Randomization coding tables will be hidden from the investigator till the end of the study.

Group I (dilation group): in which mechanical cervical dilatation will be done.

Group II (Non-dilation group): in which no mechanical cervical dilatation will be done. ***** ***Study procedure:

After taking informed written consent, the recruited patients will be subjected to the following:

Clinical examination:

* History: personal (age, duration of marriage), present (any current medical or surgical diseases and any current medication), Past (history of any medical disorder) and obstetric history (including Parity, Gestational age, obstetric complications). Indications for cesarean were determined as malposition of the fetal head, head-pelvis incompatibility, disrupted fetal heart rate.
* General examination: assessment of body mass index (BMI) ,vital data (pulse, blood pressure, temperature), cardiac and chest auscultation to exclude contraindications for anesthesia.
* Abdominal examination: assessment of fundal level, fetal lie and presentation liquor volume and previous scar if present.
* Vaginal examination: to exclude cervical changes.
* Ultrasound examination: to assess fetal viability, determine gestational age and exclude major anomalies.

Steps:

* Informed consent will be obtained from women who will be invited to participate in the research after an explanation of the benefits and risks of this trial.
* All caesarean sections will be performed by a senior registrar capable of doing uncomplicated elective cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

Elective Cs (primary or repeated CS)

Exclusion Criteria:

Medical or obstetric conditions that may put them at risk for uterine atony and postpartum hemorrhage and infection, such as:

* Emergency Cesarean section
* Chorioamnionitis.
* Preterm caesarean section.
* Multiple gestations.
* Fever during admission.
* Rupture of membranes.
* Anemia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
postpartum 6th month scar thickness | 6 months after delivery
  measure the thickness of the residual myometrial tissue (RMT) in mm by transvaginal ultrsound

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR